CLINICAL TRIAL: NCT00942643
Title: Endothelial Damage and Atherosclerosis in Obstructive Sleep Apnea: the Role of Advanced Glycation End-products
Brief Title: Endothelial Damage and Atherosclerosis in Obstructive Sleep Apnea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor patient recruitment
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lam Jamie Chung Mei, Honorary clinical assistant professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HKCTR-772
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Obstructive Sleep Apnea; Insulin Resistance; Endothelial Function; Oxidative Stress
MeSH Terms: conditions — Sleep Apnea, Obstructive; Insulin Resistance | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no treatment (No Intervention): being observed at 4 weeks and 12 weeks
- CPAP treatment (Active Comparator): a machine delivers positive airway pressure into the upper airway via nasal mask
  Interventions: Device: CPAP machine

INTERVENTIONS:
Device: CPAP machine — a machine delivers positive airway pressure into the upper airway via a nasal mask
  Other Names: Continuous Positive Airway Pressure
  Arms: CPAP treatment

SUMMARY:
The investigators hypothesize that obstructive sleep apnea (OSA) may lead to increased formation/accumulation of advanced glycation ends (AGEs), and that the increase in AGEs is contributed in part by increased insulin resistance. The investigators further hypothesize that AGEs contribute to vascular endothelial damage and ultimately atherosclerosis in OSA.

The objectives of this study are:

1. To explore the relationship between insulin resistance and AGEs in OSA
2. To study the relationship between AGE and vascular endothelial dysfunction in OSA
3. To study the relationship between AGE and early atherosclerosis in OSA

DETAILED DESCRIPTION:
There is growing evidence to suggest that pathophysiology of OSA may lead to atherosclerosis, independent of confounding variables which are often present in these subjects with OSA. Many mechanisms have been reported to contribute to vasculopathy in OSA, but whether increased AGEs formation contribute significantly to the pathogenesis of cardiovascular morbidity in OSA remains to be determined.

Advanced glycation product is formed by non-enzymatic reaction of reducing sugars such as glucose with the amino groups of proteins, and subsequent glycoxidation. AGEs can form on long-lived extracellular proteins as well as short-lived molecules, cytoplasmic proteins and nuclear acids. AGEs cause a number of adverse cellular events and they have been demonstrated in fatty streaks and atherosclerotic plaques. The formation and tissue accumulation of AGE is shown to be enhanced by hyperglycemia and/or increased oxidative stress. There is increasing evidence to support this as an important mechanism of vascular and other end organ damage in diabetes and some other diseases. In OSA, there is evidence to support an increased insulin resistance and excessive oxidative stress, both of which may predispose to AGE formation. We have preliminary data to suggest increased levels of circulating AGE in non-diabetic OSA subjects. Since insulin resistance with elevated blood glucose levels, albeit not up to diabetic thresholds, may partially contribute to increase in AGE.

Many potential mechanisms of atherosclerosis have been reported, but direct evidence for atherosclerosis is still lacking. Subjects with OSA also have comorbidities which may give rise to atherosclerosis. With the advancement of non-invasive techniques for detection of vascular endothelial damage and early atherosclerosis, it is possible to detect early vascular abnormalities in otherwise healthy OSA subjects. This hypothesis underlies our objectives to explore the relationship between AGE and the markers of endothelial dysfunction and early atherosclerosis. Some of these early changes, especially at endothelial level, may be reversible if the insult of OSA is removed. Thus a longitudinal comparison of OSA-treated and OSA-untreated subjects on such changes would further help to clarify the issue.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 years old
* AHI >= 15
* BMI < 35

Exclusion Criteria:

* Known cardiovascular disease, including hypertension
* Diabetes
* Acute or unstable chronic disease
* Renal failure
* Major organ system failure, including liver, renal, cardiac and respiratory failure
* Taking long-term medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
AGEs levels | 4 weeks and 12 weeks

SECONDARY OUTCOMES:
endothelial function as assessed by reactive hyperemia-induced peripheral arterial tone response | 4 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary SM Ip, MD, Principal Investigator — Queen Mary Hospital, The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Pokfulam, Pokfulam, Hong Kong